CLINICAL TRIAL: NCT01556373
Title: Effects of Acute Systemic Inflammation on Arterial Stiffness and Microcirculation.
Acronym: IRIGA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A00612-37
Record Dates: First submitted 2012-02-23; First posted 2012-03-16 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Severe Sepsis
Keywords: acute systemic inflammation; arterial stiffness; Carotid-femoral pulse wave velocity
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- severe sepsis: patients with severe sepsis
  Interventions: Other: NA : non interventional study
- Controls: Controls matched to patients on age, sex and cardiovascular risk factors
  Interventions: Other: NA : non interventional study

INTERVENTIONS:
Other: NA : non interventional study — NA : non interventional study

SUMMARY:
This study aims to assess the effect of acute inflammation on arterial stiffness and microcirculation. Patients with severe sepsis will be compared with age-, sex- and cardiovascular risk factors-matched controls.

The primary outcome is the carotid-femoral pulse wave velocity. The other outcome measures are: systemic hemodynamics (systolic, diastolic, mean and pulse blood pressures, heart rate, cardiac output, left ventricular ejection fraction, systemic vascular resistances), central hemodynamics (aortic systolic, diastolic, mean and pulse pressures, and augmentation index), thenar tissue oxygen saturation, biological makers of inflammation (plasma fibrinogen, C-reactive protein, interleukin-6, matrix metalloproteinases -2, -9, tissue inhibitor of metalloproteinase 1), and plasma catecholamine concentrations (epinephrine, norepinephrine).

DETAILED DESCRIPTION:
In a model of acute inflammation induced by salmonella typhi vaccination in healthy volunteers, it has been shown that acute systemic inflammation increased arterial stiffness. Since increased arterial stiffness (assessed by carotid-femoral pulse wave velocity) is an independent prognosis marker of cardiovascular risk in many chronic diseases such as hypertension, renal failure or diabetes mellitus, it could also be a marker of severity in acute inflammation states. Severe sepsis is a leading cause of hospitalisation in intensive care units, and constitutes a state of acute inflammation. It remains however to confirm that arterial stiffness is increased in this clinical conditions before evaluating its prognosis value.

This study aims to assess the effect of severe sepsis on arterial stiffness and microcirculation. Patients with severe sepsis will be compared with age-, sex- and cardiovascular risk factors-matched controls.

The primary outcome is the carotid-femoral pulse wave velocity. The other outcome measures are: systemic hemodynamics (systolic, diastolic, mean and pulse blood pressures, heart rate, cardiac output, left ventricular ejection fraction, systemic vascular resistances), central hemodynamics (aortic systolic, diastolic, mean and pulse pressures, and augmentation index), thenar tissue oxygen saturation, biological makers of inflammation (plasma fibrinogen, C-reactive protein, interleukin-6, matrix metalloproteinases -2, -9, tissue inhibitor of metalloproteinase 1), and plasma catecholamine concentrations (epinephrine, norepinephrine).

ELIGIBILITY:
Inclusion Criteria:

* Control group :

  * male or female aged at least 18 years, matched on age, sex and cardiovascular risk factors (smoking, hypertension, diabetes and treated dyslipidemia) with septic patients
  * Normal clinical examination and normal 12-lead ECG
  * Routines biological tests in the normal range of the laboratories.
  * Body mass index between 18 and 27 kg/m²
  * Written informed consent
* Patients group :

  * Male or female aged at least 18 years
  * Severe sepsis defined by the presence of:

    * a systemic inflammatory response syndrome
    * the evidence of an infection
    * the presence of at least one organ failure or signs of tissue hypoperfusion.
  * Body mass index between 18 and 27 Kg/m²
  * Written informed consent from the patients or their relatives

Exclusion Criteria:

* Control group :

  * legal protection or persons deprived of liberty
  * bacterial or viral infection in the month preceding inclusion
  * current medication
  * pregnancy or breastfeeding
  * exclusion period stated on the national register for persons who participate to biomedical research
* Patients group :

  * legal protection or persons deprived of liberty
  * vasopressor therapy
  * bacterial or viral infection in the month preceding inclusion
  * known cardiomyopathy
  * pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with severe sepsis. 20 controls matched on age, sex and cardiovascular risk factors .
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral pulse wave velocity | 1 day

SECONDARY OUTCOMES:
Systemic hemodynamics | 1 day
  * Systolic, diastolic, mean, and pulse blood pressures, and heart rate
  * Cardiac output, left ventricular ejection fraction, systemic vascular resistances
Central aortic hemodynamic | 1 day
  * Aortic systolic, diastolic, mean and pulse pressures,
  * Augmentation index
Micro-circulation | 1 day
  Thenar tissue oxygen saturation
Biological markers from plasma samples | 1 day
  * fibrinogen
  * C-reactiv protein
  * Interleukin-6
  * matrix metalloproteinases -2, -9, and tissue inhibitor of metalloproteinase 1
  * epinephrine and norepinephrine

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LAVIOLLE, MD, PhD, Principal Investigator — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (2):
- France (2):
  - Service de Réanimation Chirurgicale - Hôpital de Pontchaillou, Rennes
  - Unité d'Investigation Clinique - Hôpital de Pontchaillou, Rennes